CLINICAL TRIAL: NCT01331291
Title: An Open Label, Phase 2 Trial of Orally Administered Bosutinib (SKI-606) in Adult Patients With Recurrent Glioblastoma (GBM)
Brief Title: Bosutinib in Adult Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Tracy T. Batchelor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-190
Record Dates: First submitted 2011-03-28; First posted 2011-04-08 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Glioblastoma
Keywords: bosutinib; SKI-606
MeSH Terms: conditions — Glioblastoma | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients who are surgical candidates. Participants are given oral bosutinib, 400mg daily, for 7-9 days prior to resection. After at least 10 days elapsed post-operatively, bosutinib dosing was resumed.
  Interventions: Drug: bosutinib
- Arm B (Experimental): Patients that are not surgical candidates. Participants are given oral bosutinib, 400 mg daily in 28 day cycles until disease progression, intolerability or withdrawal of consent.
  Interventions: Drug: bosutinib

INTERVENTIONS:
Drug: bosutinib — Taken orally
  Other Names: SKI-606

SUMMARY:
For many brain tumors, one reason that chemotherapy drugs might not be effective is that the drug may not be able to get into the brain tumor and kill the cancer cells. The brain is protected by a layer called the blood brain barrier. This barrier prevents substances from entering. The purpose of this research study is to determine if bosutinib can get past the blood brain barrier and into the brain tumor, and to see how well bosutinib works in killing cancer cells.

DETAILED DESCRIPTION:
- Arm A: Participants will receive daily doses of bosutinib orally for 7-9 days prior to surgery. On the day of the scheduled surgery (either craniotomy or surgical resection as planned by the treating doctor), participants will take the bosutinib within 6-12 hours of the surgery. During the surgery, tissue samples of the tumor will be collected to test the levels of bosutinib in the brain. A contrast-enhanced MRI or CT scan will be done within days after the surgery. Daily dosing of bosutinib will resume after a recovery period of 10 days. From then on, the study will be divided into 28-day cycles.

The following tests/procedures will be performed regularly during cycles of study treatment: medical history; physical exam; blood tests; contrast-enhanced CT or MRI scans (even numbered cycles only).

* Arm B: Participants will receive daily doses of bosutinib. The study is divided int 28-day cycles. There are no breaks from taking bosutinib between treatment cycles. The following tests/procedures will be performed regularly during cycles of study treatment: medical history; physical exam; blood tests; contrast-enhanced CT or MRI scans (even numbered cycles only).
* Participants may continue to receive daily bosutinib until their disease worsens, they experience unmanageable side-effects, or they decide to stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed WHO (World Health Organization) grade IV astrocytoma (glioblastoma). Patients with recurrent disease whose original pathology confirmed glioblastoma will not need re-biopsy. Patients with prior low-grade glioma or anaplastic glioma are eligible if histological assessment demonstrates transformation to GBM.
* The first-line regimen must have included, at a minimum, temozolomide and radiation.
* First or second episode of progressive disease.
* No more than two prior treatment regimens for progressive disease. Concurrent temozolomide and radiation followed by monthly cycles of temozolomide is counted as one regimen.
* For all study arms, patients must have at least 15 unstained slides or 1 tissue block available from a prior biopsy or surgery.
* All patients must have progressive disease on contrast-enhanced brain CT or MRI as defined by MacDonald Criteria, or have documented recurrent glioblastoma on diagnostic biopsy. Arm A patients may continue treatment in the post-operative period even if there is no residual contrast-enhancing tumor after surgery.
* For Arm A, patients must be candidates for surgical partial or gross-total resection.
* Interval of at least 2 weeks between prior surgical resection and adequate wound healing.
* Interval of at least 12 weeks from prior radiotherapy unless there is either a) histopathologic confirmation of recurrent tumor; b) new enhancement on MRI outside of the XRT (external beam radiation therapy) treatment field.
* Patients must have sufficient time for recovery from prior therapy
* Karnofsky Performance Status of 60% or greater
* Laboratory levels as outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months thereafter.

Exclusion Criteria:

* Participants may not be receiving any other investigational agents
* Previously treated with an anti-VEGF (anti-vascular endothelial growth factor) agent
* For subjects in Arm A: if the diagnostic pathology of the biopsy specimen is not consistent with recurrent glioblastoma then the subject will be taken off study and be replaced with another subject that meets the inclusion criteria and is eligible for surgical resection
* Any surgery within 2 weeks of baseline disease assessments, or not fully recovered from any side effects of previous procedures
* Any clinically significant gastrointestinal abnormalities, which may impair intake, transit or absorption of the study drug, such as the inability to take oral medications in tablet form.
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this protocol
* Concomitant use of CYP3A4/5 inhibitors during the treatment phase of the study and within 72 hours prior to starting study drug administration
* Concomitant use of CYP3A4/5 inducers, which include enzyme inducing antiepileptic drugs during treatment phase of the study and within 2 weeks prior to starting treatment.
* Uncontrolled or significant cardiovascular disease
* Prior stereotactic radiotherapy, convection enhanced delivery or brachytherapy as gliosis/scarring from these modalities may limit delivery
* Pregnant or breast feeding women
* HIV-positive individuals on combination antiretroviral therapy
* Other severe acute or chronic medical condition or laboratory abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana=Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taylor JW, Dietrich J, Gerstner ER, Norden AD, Rinne ML, Cahill DP, Stemmer-Rachamimov A, Wen PY, Betensky RA, Giorgio DH, Snodgrass K, Randall AE, Batchelor TT, Chi AS. Phase 2 study of bosutinib, a Src inhibitor, in adults with recurrent glioblastoma. J Neurooncol. 2015 Feb;121(3):557-63. doi: 10.1007/s11060-014-1667-z. Epub 2014 Nov 20. PMID 25411098

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Patients who are surgical candidates
  bosutinib: Taken orally
- Arm B: Patients that are not surgical candidates
  bosutinib: Taken orally
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 2 | 9
Completed | 0 | 0
Not Completed | 2 | 9
Not completed — Lack of Efficacy | 2 | 8
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 2 | 9 | 11
Age, Continuous [Median (Full Range); unit: years] | 60 [58 to 62] | 44 [36 to 62] | 52 [36 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 2 | 5 | 7
Prior Surgery [Number; unit: participants] — Surgery done at time of diagnosis with glioblastoma
  participants
    Gross Total Resection | 1 | 6 | 7
    Sub total Resection | 0 | 3 | 3
    No prior surgery | 1 | 0 | 1
Karnofsky Performance Status (KPS) [Median (Full Range); unit: units on a scale] — A standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. (0 being 'Dead' and 100 being 'Normal, no complaints; no evidence of disease'.)
  units on a scale | 80 [70 to 90] | 90 [70 to 90] | 90 [70 to 90]
Prior chemoradiation [Number; unit: participants] — Number of patients who previously received standard, initial therapy with temozolomide and radiation at diagnosis
  participants | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Assess progression-free survival at six months in patients with recurrent glioblastoma at first or second recurrence who are treated with continuous daily dosing of bosutinib (Arm B). Progression-free survival is measured from initiation of study treatment to date of progression.
Time Frame: 2 years
Population: This outcome was only applicable to participants enrolled on Arm B.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 9
weeks |  | 7.71 [2.6 to 7.9]

2. Secondary Outcome: Intratumoral Concentration
Description: Assess the intratumoral concentration of bosutinib in recurrent glioblastoma patients who are candidates for surgical re-resection (ARM A).
Time Frame: 2 years
Population: Participants in Arm B were never eligible for this outcome measure. Because only two participants were enrolled to Arm A, this analysis was not done as there were not sufficient tumor samples to generate meaningful results.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Safety Profile
Description: Overall safety profile will be characterized by type, frequency, severity (as graded by NCI CTCAE), timing and relationship of study therapy of adverse events and laboratory abnormalities. Safety and tolerability will be measured by the proportion of patients who experience Grade 3 or higher Adverse Events that are possibly, probably or definitely related to bosutinib and the number of same Adverse Events per patient. Adverse Events will be summarized by treatment for each arm by the frequency of patients experiencing treatment emergent adverse events.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 9
participants
  Grade 3 treatment-emergent lymphopenia | 0 | 1
  Grade 3 treatment-emergent hypophosphatemia | 0 | 1

4. Secondary Outcome: Anti-tumor Response
Description: Assess anti-tumor response in patients in Arm B using MacDonald criteria. There are four possible responses: complete response, partial response, stable disease, or progressive disease. Criteria are based on measurements of tumor dimension as visualized with a contrast-enhanced MRI.
Time Frame: 2 years
Population: Only Arm B participants were evaluable for this outcome measure
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 9
participants
  Complete response |  | 0
  Partial response |  | 0
  Stable Disease |  | 1
  Progressive disease |  | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were followed for the duration of the participants' time on study; an average of two 28-day cycles (56 total days), with a range of one to six cycles.
Groups:
- Combined Arms: Adverse Events were measured across all participants, regardless of arm.
Arm/Group | Combined Arms
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Arms (N=11)
cellulitis (Skin and subcutaneous tissue disorders) | 1
seizure (Nervous system disorders) | 1
fall (Injury, poisoning and procedural complications) | 1
lymphocyte count decreased (Investigations) | 1
lung infection (Infections and infestations) | 1
diarrhea (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
dizziness (Nervous system disorders) | 1
vomiting (Gastrointestinal disorders) | 1
headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Arms (N=11)
lymphocyte count decreased (Investigations) | 8
fatigue (General disorders) | 6
nausea (Gastrointestinal disorders) | 5
seizure (Nervous system disorders) | 4
elevated alanine aminotransferase (Investigations) | 5
diarrhea (Gastrointestinal disorders) | 3
hypophosphatemia (Metabolism and nutrition disorders) | 4
rash (Skin and subcutaneous tissue disorders) | 3
lung infection (Infections and infestations) | 2
elevated aspartate aminotransferase (Investigations) | 2
cerebral edema (Nervous system disorders) | 1
maculo-papular rash (Skin and subcutaneous tissue disorders) | 4

LIMITATIONS AND CAVEATS:
This study met pre-specified criteria for early closure, as all 9 patients enrolled on Arm B demonstrated disease progression within 6 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No